CLINICAL TRIAL: NCT02763228
Title: A Physical Activity Intervention to Reduce Functional Health Disparities Among Older Breast Cancer Survivors
Brief Title: Physical Activity Intervention to Reduce Functional Health Disparities Among Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE2116
Record Dates: First submitted 2016-04-27; First posted 2016-05-05 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer; Physical Activity
Keywords: Physical Activity; Breast Cancer; minority; African American
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise; Self-Help Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Exercise Program (Experimental): The exercise in this study will consist of two types of exercise training: resistance training and aerobic exercise. Resistance training is like "weight lifting" to improve strength and function. Participants will complete resistance training by using resistance machines and free weights. Aerobic exercise is exercise that intends to improve the cardiopulmonary or oxygen/lung and heart systems. It is often referred to as "cardio" exercise. Treadmill walking, stationary cycling sessions, and/or other exercises will be used for aerobic exercise.
  Participants will be instructed in the exercise routine by physical fitness experts and trainers.
  Interventions: Behavioral: Aerobic Training - Fixed Schedule; Behavioral: Resistance Training - Fixed Schedule; Behavioral: Walking program; Behavioral: Aerobic Training - Flexible Schedule; Behavioral: Resistance Training - Flexible Schedule
- Group 2: Support Group (Active Comparator): First 20 Weeks: Participants will take part in a structured Health Education and Support Group sessions once a week.
  Last 32 weeks: Participants will be encouraged to take part in any of the Support Group sessions offered regularly on their own schedule.
  Interventions: Behavioral: Successful Survivorship Health Education and Support Group; Behavioral: Flexible support groups

INTERVENTIONS:
Behavioral: Aerobic Training - Fixed Schedule — Supervised aerobic training for 40 minutes 3x/week for 20 weeks
  Other Names: Aerobic exercise
  Arms: Group 1: Exercise Program
Behavioral: Resistance Training - Fixed Schedule — Supervised resistance training for 20 minutes 3x/week for 20 weeks
  Arms: Group 1: Exercise Program
Behavioral: Walking program — Unsupervised walking program 1-3 days/week for 52 weeks
  Arms: Group 1: Exercise Program
Behavioral: Aerobic Training - Flexible Schedule — Supervised aerobic training done on the participant's own schedule for 32 weeks
  Arms: Group 1: Exercise Program
Behavioral: Resistance Training - Flexible Schedule — Supervised resistance training done on the participant's own schedule for 32 weeks
  Arms: Group 1: Exercise Program
Behavioral: Successful Survivorship Health Education and Support Group — Support groups will be held for one hour 3x/week for 20 weeks. Topics will include, but are not limited, to long-term side effects of treatment, stress management, coping with fear and uncertainty, body image, sexuality, and spirituality.
  Other Names: Structured Support Group
  Arms: Group 2: Support Group
Behavioral: Flexible support groups — Participants will attend 1-3 weekly group sessions of their choosing for 32 weeks.
  Arms: Group 2: Support Group

SUMMARY:
The purpose of this research study is to determine whether a physical activity (exercise) program in the community will improve the functional and overall health status of older women with a history of breast cancer. The physical activity or exercise program is designed for all older breast cancer survivors, and in particular for African-Americans and women of lower socio-economic status, who are the least likely to engage in physical activity.

DETAILED DESCRIPTION:
Specific Aim #1: To determine the effect of a refined and culturally-sensitive physical activity intervention on functional outcomes at 20 and 52 weeks among older Breast Cancer survivors who are within five years of treatment completion for stage I-III Breast Cancer (BCa).

Specific Aim #2: To examine whether race and socioeconomic status (SES) moderate the intervention effect on physical activity (PA) levels and functional outcomes at 20 and 52 weeks.

Specific Aim #3: To examine the effect of the PA intervention on longitudinal changes in beliefs, attitudes and preferences (KAPs) and PA levels, and the extent to which changes in these factors mediate intervention effect on functional outcomes.

Specific Aim #4: To determine the effect of the PA intervention on surrogate biomarkers associated with breast cancer prognosis and functional disability.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed breast cancer
* Stage I-III
* Patients who have completed treatment but are within five years of treatment completion (primary surgery, chemotherapy or radiation therapy), whichever was received last. Hormonal therapy and targeted therapy are allowed
* Race: African-Americans and Non-Hispanic Whites

Exclusion Criteria:

* Stage IV breast cancer
* Patients with end-stage disease, severe dementia and/or life expectancy of less than one year
* Inability to understand English as study instruments have not been validated in other languages
* Inability to provide informed consent
* High-risk patients (as defined by the American College of Sports Medicine risk-stratification schema using the American College of Sports Medicine (ACSM)/American Heart Association exercise pre-participation questionnaire) who do not receive clearance from cardiology
* Other medical or psychological conditions that would make participation unsafe or inhibit our ability to test our primary hypothesis, e.g. Parkinson's disease, severe dementia.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 218 (Actual)
Dates: Start 2016-03-16 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
Change in physical performance scores based on the Short Physical Performance Battery (SPPB) | baseline to 20 weeks
  Change in physical performance will be ascertained using the Short Physical Performance Battery (SPPB). Summary scores range from 0-12 and higher scores denote higher physical performance.

SECONDARY OUTCOMES:
Change in SPPB scores | baseline to 52 weeks
  Change in physical performance will be ascertained using the Short Physical Performance Battery (SPPB). Summary scores range from 0-12 and higher scores denote higher physical performance.
Change in Activities of daily living (ADL) score | baseline to 20 weeks
  Summary scores for ADL range from 0-14 and higher scores denote higher functional status.
Change in Activities of daily living (ADL) score | baseline to 52 weeks
  Summary scores for ADL range from 0-14 and higher scores denote higher functional status.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Owusu, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Metro Health Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center, Cleveland, Ohio

REFERENCES:
- [Derived] Hundal J, Williams D, Nock NL, Austin K, Bennet E, Cerne S, Moore HCF, Petkac J, Schmitz KH, Berger NA, Owusu C. Older breast cancer survivors' exercise and support group program experiences and recommendations from the IMPROVE trial: a qualitative study. BMC Cancer. 2026 Jan 6;26(1):181. doi: 10.1186/s12885-025-15425-w. PMID 41495697
- [Derived] Owusu C, Margevicius S, Nock NL, Austin K, Bennet E, Cerne S, Hergenroeder P, Moore HCF, Petkac J, Schluchter M, Schmitz KH, Webb Hooper M, Wimbley L, Berger NA. A randomized controlled trial of the effect of supervised exercise on functional outcomes in older African American and non-Hispanic White breast cancer survivors: Are there racial differences in the effects of exercise on functional outcomes? Cancer. 2022 Jun 15;128(12):2320-2338. doi: 10.1002/cncr.34184. Epub 2022 Mar 15. PMID 35289926
- [Derived] Owusu C, Nock NL, Feuntes V, Margevicius S, Hergenroeder P, Austin K, Bennet E, Cerne S, Moore HCF, Petkac J, Schluchter M, Schmitz KH, Webb Hooper M, Coccia S, Nagy C, Wimbley L, Berger NA. IMPROVE, a community-based exercise intervention versus support group to improve functional and health outcomes among older African American and Non-Hispanic White breast cancer survivors from diverse socioeconomic backgrounds: Recruitment strategies and baseline characteristics. Cancer. 2021 Jun 1;127(11):1836-1846. doi: 10.1002/cncr.33430. Epub 2021 Feb 4. PMID 33539554